CLINICAL TRIAL: NCT05356312
Title: Retrospective Analysis of Glioblastoma Patients With Immune Therapies
Brief Title: Glioblastoma and Individualized Therapies
Status: Available | Type: Expanded Access
Sponsor: Zentrum fur Humangenetik Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: GBM-RWD
Record Dates: First submitted 2022-04-11; First posted 2022-05-02 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Glioma, Malignant
MeSH Terms: conditions — Glioma | interventions — Vaccination

INTERVENTIONS:
Biological: Vaccination — Personalized neoantigen vaccination

SUMMARY:
The treatment of patients with World Health Organization (WHO) grade 4 malignant glioma has not seen any significant breakthrough the past years. Following surgery and radio / chemotherapy patients still experience a very high recurrence risk and the prognosis is dismal. The investigators observed patients with grade IV malignant glioma receiving individualized treatment based on their molecular profile including fully personalized vaccines.

ELIGIBILITY:
Inclusion Criteria:

* malignant glioma, IDH WT

Exclusion Criteria:

* na

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Zentrum für Humangenetik Tübingen, Tübingen, Germany